CLINICAL TRIAL: NCT04513366
Title: A Randomized Double-Blind, Placebo-Controlled Study of SEL-212 in Patients With Gout Refractory to Conventional Therapy
Brief Title: A Study of SEL-212 in Patients With Gout Refractory to Conventional Therapy
Acronym: DISSOLVE I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SEL-212/301
Record Dates: First submitted 2020-08-07; First posted 2020-08-14 (Actual); Results first posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Chronic Gout
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SEL-212 low-dose (Experimental): SEL-212 low-dose Drug: SEL-037 (0.2 mg/kg) SEL-037, PEGylated uric acid specific enzyme (uricase)
  Other Names:
  Pegadricase, pegsiticase Drug: SEL-110.36 (0.1 mg/kg) SEL-110.36, ImmTOR
  Interventions: Drug: SEL-212 low-dose
- SEL-212 high-dose (Experimental): SEL-212 high-dose Drug: SEL-037 (0.2 mg/kg) SEL-037, PEGylated uric acid specific enzyme (uricase)
  Other Names:
  Pegadricase, pegsiticase Drug: SEL-110.36 (0.15 mg/kg) SEL-110.36, ImmTOR
  Interventions: Drug: SEL-212 high-dose
- Placebo (Placebo Comparator): Normal saline
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: SEL-212 low-dose — IV infusion of SEL-212 low-dose every 28 days for a total of up to 12 infusions
  Arms: SEL-212 low-dose
Drug: SEL-212 high-dose — IV infusion of SEL-212 high-dose every 28 days for a total of up to 12 infusions
  Arms: SEL-212 high-dose
Other: Normal Saline — IV infusion of Normal Saline every 28 days for a total of up to 12 infusions
  Arms: Placebo

SUMMARY:
This is one of two replicate randomized, double-blind, placebo-controlled, parallel arm trials to determine the safety and efficacy of two different dose levels of SEL-212 compared to placebo. 112 and 153 patients, stratified as to the presence or absence of tophi, were randomized in a 1:1:1 allocation ratio prior to Baseline to receive treatment with one of two dose levels of SEL-212 or placebo every 28 days for approximately 6 months in each trial respectively (SEL-212/301 and SEL-212/302). Analysis of primary and key efficacy was performed at Day 28 of Treatment Period 6. Safety was monitored throughout the study.

DETAILED DESCRIPTION:
This is one of two replicate randomized, double-blind, placebo-controlled, parallel arm trials to determine the safety and efficacy of two different dose levels of SEL-212 compared to placebo. 112 and 153 patients, stratified as to the presence or absence of tophi, were randomized in a 1:1:1 allocation ratio prior to Baseline to receive treatment with one of two dose levels of SEL-212 or placebo every 28 days for approximately 6 months in each trial respectively (SEL-212/301 and SEL-212/302). The SEL-212 doses differed as to the SEL-110.36 component. Participants received SEL-037 administered at a dose of 0.2 mg/kg via intravenous (IV) infusion immediately after receiving SEL-110.36 at a dose of either 0.1 mg/kg (SEL-212 low-dose) or 0.15 mg/kg (SEL-212 high-dose) via IV infusion. The placebo consisted of normal saline.

Upon completion of the 6-month double-blinded, placebo-controlled portion of the study, SEL-212/301 continued in a blinded, placebo-controlled 6-month extension. This provided up to 12 months of continuous treatment with SEL-212 in a placebo controlled fashion.

Efficacy assessments were conducted at intervals that are appropriate to determine treatment effect with samples for the primary endpoint drawn during Treatment Period 6. Safety was monitored throughout the study with an independent data safety monitoring board (DSMB).

ELIGIBILITY:
Inclusion Criteria:

1. Has negative results of an FDA Emergency Use Authorized COVID-19 molecular assay for detection of SARS-CoV-2 RNA from a nasal or oropharyngeal specimen;
2. History of symptomatic gout defined as:

   1. ≥ 3 gout flares within 18 months of Screening or
   2. Presence of ≥ 1 gout tophus or
   3. Current diagnosis of gouty arthritis
3. At the Screening Visit: male age 21 - 80 years, inclusive, or female of non-childbearing potential age 21-80 years, inclusive, where nonchildbearing potential is defined as:

   a. > 6 weeks after hysterectomy with or without surgical bilateral salpingooperhectony or b. Post-menopausal (> 24 months of natural amenorrhea or in the absence of >24 months of amenorrhea, one documented confirmatory FSH measurement)
4. Has chronic refractory gout defined as having failed to normalize sUA and whose signs and symptoms are inadequately controlled with any of the xanthine oxidase inhibitors, or for whom these drugs are contraindicated for the patient;
5. Has at the Screening Visit SUA ≥ 7 mg/dL
6. Negative serology for HIV-1/-2 and negative antigen to hepatitis B and negative antibodies to hepatitis C;

Exclusion Criteria:

1. Has a history of anaphylaxis, severe allergic reactions, or severe atopy;
2. Has a history of any allergy to pegylated products, including, but not limited to pegloticase (Krystexxa®), peginterferon alfa-2a (Pegasys®), peginterferon alfa-2b (PegIntron®), pegfilgrastim (Neulasta®), pegaptanib (Macugen®), pegaspargase (Oncaspar®), pegademase (Adagen®), peg-epoetin beta (Mircera®), pegvisomant (Somavert®) certolizumab pegol (Cimzia®), naloxegol (Movantik®), peginesatide (Omontys®), and doxorubicin liposome (Doxil®);
3. Is taking and cannot discontinue known major CYP3A4/P-gp inhibitors or major CYP3A4/P-gp inducers at least 14 days before dosing. Patients must remain off these medications for the duration of the study, including natural products such as St. John's Wort or grapefruit juice.
4. Is taking drugs known to interact with rapamycin (sirolimus - Rapamune®) such as cyclosporine, diltiazem, erythromycin, ketoconazole, posaconazole, voriconazole, itraconazole, rifampin, verapamil unless they are stopped 14 days prior to dosing and will not be used/prescribed during the trial.
5. Had major surgery within 3 months of initial screening.
6. Had a gout flare during Screening that was resolved for less than 1 week prior to first treatment with study drug (exclusive of chronic synovitis/arthritis) unless the patient has a history of inter-flare intervals of < 1 week.
7. Has uncontrolled diabetes at Screening with HbA1c ≥ 8.5%;
8. Has fasting Screening glucose > 240 mg/dL;
9. Has fasting Screening triglyceride > 500 mg/dL;
10. Has fasting Screening low-density lipoprotein (LDL) > 200 mg/dL;
11. Has glucose-6-phosphate dehydrogenase (G6PD) deficiency;
12. Has uncontrolled hypertension defined as blood pressure > 170/100 mmHg at Screening and 1 week prior to dosing
13. Individual laboratory values which are exclusionary

    * White blood cell count (WBC) < 3.0 x109/L
    * Serum aspartate aminotransferase (AST) or alanine amino transferase (ALT) > 3x upper limit of normal (ULN) in the absence of known active liver disease
    * Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2
    * Urine albumin creatinine ratio (UACR) > 30 mg/g
    * Hemoglobin (Hgb) < 9 g/dL
    * Serum phosphate < 2.0 mg/dL
14. Is receiving ongoing treatment for arrhythmia, including placement of an implantable defibrillator, unless considered stable and on active treatment;
15. Has evidence of unstable cardiovascular disease or unstable cerebrovascular vascular disease. This includes patients who have had a cardiac/vascular event(s) in the last 3 months including heart attack, stroke or vascular bypass surgery or patients who are deemed, by their physician or PI, to have active cardiovascular, cerebrovascular or peripheral vascular symptoms/disease inadequately controlled by medication;
16. Has congestive heart failure, New York Heart Association Class III or IV;
17. Unless clinically stable and/or appropriately treated, electrocardiogram (ECG) with evidence of clinically significant arrhythmia or other abnormalities that, in the opinion of the investigator, are consistent with significant underlying cardiac disease;
18. History of significant hematological disorders within 5 years or autoimmune disorders, and/or patient is currently immunosuppressed or immunocompromised;
19. Prior exposure to any experimental or marketed uricase (e.g., rasburicase (Elitek, Fasturtec), pegloticase (Krystexxa®), pegadricase (SEL 37))
20. Patient has received a live vaccine in the previous 6 months.
21. Patient is planning to receive any live vaccine during the study.
22. History of malignancy within the last 5 years other than basal skin cancer;
23. Patients with a documented history of moderate or severe alcohol or substance use disorder within the 12 months prior to randomization.
24. History of or evidence of clinically severe interstitial lung disease
25. Immunocompromised state, regardless of etiology

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female of non-childbearing potential defined as either >6 weeks after hysterectomy with or without surgical bilateral salpingo-oophorectomy OR post-menopausal (> 24 months of natural amenorrhea or in the absence of > 24 months of amenorrhea, one documented confirmatory FSH measurement)
Enrollment: 112 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (40):
- United States (40):
  - Pinnacle Research Group, Anniston, Alabama
  - Arizona Arthritis & Rheumatology Research, PLLC, Sun City, Arizona
  - Medvin Clinical Research, Covina, California
  - Valerius Medical Group & Research Center, Los Alamitos, California
  - ACRC Studies, Poway, California
  - MD Strategies Research Center, San Diego, California
  - Tekton Research - Fort Collins, Fort Collins, Colorado
  - Helix Biomedics, LLC, Boynton Beach, Florida
  - Clinical Research Of West Florida Incorporated, Clearwater, Florida
  - Omegas Research Consultants LLC, DeBary, Florida
  - Riverside Clinical Research, Edgewater, Florida
  - Homestead Associates in Research,Inc, Homestead, Florida
  - Health Awareness INC, Jupiter, Florida
  - Y & L Advance Health Care, Inc, Miami, Florida
  - Well Pharma Medical Research, Corp, Miami, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Conquest Research, Winter Park, Florida
  - Better Health Clinical Research, Inc., Newnan, Georgia
  - Institute of Arthritis Research, Idaho Falls, Idaho
  - Advanced Clinical Research (ACR) - Family Practice/General Medicine - Meridian, Meridian, Idaho
  - L-MARC Research Center, Louisville, Kentucky
  - Research Integrity, LLC, Owensboro, Kentucky
  - Klein and Associates, M.D., P.A., Cumberland, Maryland
  - Klein and Associates, M.D., P.A., Hagerstown, Maryland
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Elite Clinical Research, LLC, Jackson, Mississippi
  - Arthritis Consultants, Inc., St Louis, Missouri
  - Montana Medical Research, Inc., Missoula, Montana
  - Medex Healthcare Research, Inc., New York, New York
  - CFA - Cape Fear Arthritis Care, PLLC, Leland, North Carolina
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Arthritis & Rheumatology Center of Oklahoma, PLLC, Oklahoma City, Oklahoma
  - West Tennessee Research Institute, Jackson, Tennessee
  - Metroplex Clinical Research Center, Dallas, Texas
  - Pioneer Research Solutions, Inc., Houston, Texas
  - Southwest Rheumatology Research LLC, Mesquite, Texas
  - AIM Trials - Internal Medicine, Plano, Texas
  - Epic Medical Research, Red Oak, Texas
  - Clinical Research Partners, LLC, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- SEL-212A (Low-dose): SEL-212 is comprised of 2 components: SEL-037 and SEL-110. Participants received SEL-037 administered at a dose of 0.2 milligrams per kilogram (mg/kg) via intravenous (IV) infusion immediately after receiving SEL-110 at a dose of 0.1 mg/kg (SEL-212A) every 28 days for approximately six months during the double-blind treatment phase.
  After completion of the double-blind treatment phase, participants continued into the double-blind extension phase. In this phase, participants continued in the identical study treatment group (SEL-212A [low-dose]) for six additional doses, every 28 days, lasting up to approximately an additional six months.
- SEL-212B (High-dose): SEL-212 is comprised of 2 components: SEL-037 and SEL-110. Participants received SEL-037 administered at a dose of 0.2 mg/kg via IV infusion immediately after receiving SEL-110 at a dose of 0.15 mg/kg (SEL-212B) every 28 days for approximately six months during the double-blind treatment phase.
  After completion of the double-blind treatment phase, participants continued into the double-blind extension phase. In this phase, participants continued in the identical study treatment group (SEL-212A [high-dose]) for six additional doses, every 28 days, lasting up to approximately an additional six months.
- Placebo: Participants received placebo (normal saline) via IV infusion every 28 days for approximately six months during the double-blind treatment phase.
  After completion of the double-blind treatment phase, participants continued into the double-blind extension phase. In this phase, participants continued in the identical study treatment group (placebo) for six additional doses, every 28 days, lasting up to approximately an additional six months.
Period: Treatment Phase
Arm/Group | SEL-212A (Low-dose) | SEL-212B (High-dose) | Placebo
Started | 37 | 38 | 37
Received at Least 1 Dose of Study Treatment | 37 | 38 | 37
Completed | 27 | 27 | 26
Not Completed | 10 | 11 | 11
Not completed — Withdrawal by Subject | 6 | 8 | 3
Not completed — Lost to Follow-up | 1 | 2 | 5
Not completed — Other than Specified | 1 | 0 | 2
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 1
Period: Extension Phase
Arm/Group | SEL-212A (Low-dose) | SEL-212B (High-dose) | Placebo
Started | 27 | 27 | 26
Received at Least 1 Dose of Study Treatment | 27 | 27 | 26
Completed | 19 | 23 | 22
Not Completed | 8 | 4 | 4
Not completed — Withdrawal by Subject | 3 | 1 | 1
Not completed — Other than Specified | 4 | 0 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Sponsor Decision | 0 | 1 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Set, which included all participants who were administered any amount of study drug. Participants were analyzed according to the treatment received.
Groups:
- Total: Total of all reporting groups
Arm/Group | SEL-212A (Low-dose) | SEL-212B (High-dose) | Placebo | Total
Number analyzed (Participants) | 37 | 38 | 37 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (10.55) | 53.6 (11.99) | 53.6 (10.57) | 54.2 (11.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 0 | 5
  Male | 35 | 35 | 37 | 107
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 6 | 10 | 30
  Not Hispanic or Latino | 23 | 32 | 27 | 82
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 0 | 3
  Black or African American | 6 | 9 | 7 | 22
  White | 28 | 27 | 22 | 77
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Who Achieved and Maintained Reduction in Serum Uric Acid (sUA) < 6 Milligrams Per Deciliter (mg/dL) for At Least 80% of The Time During Treatment Period 6 (Month 6)
Time Frame: Month 6
Population: Intent-to-Treat Set, which included all randomized and dosed participants, including participants with missing data that were multiple imputed. Participants were analyzed according to randomized treatment.
Measure: Number; unit: proportion of participants
Arm/Group | SEL-212A (Low-dose) | SEL-212B (High-dose) | Placebo
Number analyzed (Participants) | 37 | 38 | 37
proportion of participants | 0.48 | 0.56 | 0.04
Statistical Analysis 1: Comparison: SEL-212A (Low-dose) vs Placebo; Test type: Superiority; p < .0001, Mantel Haenszel; Risk Difference (RD) = 0.44, 97.5% CI 2-sided [0.23 to 0.64]
Statistical Analysis 2: Comparison: SEL-212B (High-dose) vs Placebo; Test type: Superiority; p < .0001, Mantel Haenszel; Risk Difference (RD) = 0.53, 97.5% CI 2-sided [0.32 to 0.73]

2. Secondary Outcome: Change From Baseline in Mean sUA
Time Frame: Baseline, Up to 6 months
Population: Intent-to-Treat Set, which included all randomized and dosed participants including participants with missing data that were multiple imputed. Participants were analyzed according to randomized treatment.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | SEL-212A (Low-dose) | SEL-212B (High-dose) | Placebo
Number analyzed (Participants) | 37 | 38 | 37
mg/dL | -5.1 (0.6) | -5.5 (0.6) | 0.2 (0.6)
Statistical Analysis 1: Comparison: SEL-212A (Low-dose) vs Placebo; Test type: Superiority; p < .001, ANCOVA; Least Square (LS) Mean Difference = -5.3, 97.5% CI 2-sided [-7.18 to -3.42]
Statistical Analysis 2: Comparison: SEL-212B (High-dose) vs Placebo; Test type: Superiority; p < .001, ANCOVA; LS Mean Difference = -5.6, 97.5% CI 2-sided [-7.57 to -3.70]

3. Secondary Outcome: Percentage Change From Baseline in Mean sUA
Time Frame: Baseline, Up to 6 months
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | SEL-212A (Low-dose) | SEL-212B (High-dose) | Placebo
Number analyzed (Participants) | 37 | 38 | 37
percentage change | -58.7 (8.0) | -64.2 (7.1) | 5.6 (6.8)
Statistical Analysis 1: Comparison: SEL-212A (Low-dose) vs Placebo; Test type: Superiority; p < .001, ANCOVA; LS Mean Difference = -64.3, 97.5% CI 2-sided [-87.85 to -40.85]
Statistical Analysis 2: Comparison: SEL-212B (High-dose) vs Placebo; Test type: Superiority; p < .001, ANCOVA; LS Mean Difference = -69.8, 97.5% CI 2-sided [-92.16 to -47.35]

4. Secondary Outcome: Change From Baseline in the Physical Component Summary Score of the Short Form Health Survey (SF-36)
Description: The SF-36 is a 36-item scale constructed to survey health status and quality of life (QoL). The SF-36 assesses 8 health concepts, which are the weighted sums of the questions in their section: limitations in physical activities because of health problems; limitations in social activities because of physical or emotional problems; limitations in usual role activities because of physical health problems; bodily pain; general mental health (psychological distress and well-being); limitations in usual role activities because of emotional problems; vitality (energy and fatigue); and general health perceptions. Each scale was directly transformed into a 0-100 scale, and the total average scores were calculated across the 8 health concepts. The 8 domains contributed to physical component summary and mental component summary scores. Total scores for the physical component summary score ranged from 0-100, with a higher score indicating better health outcomes.
Time Frame: Baseline, Up to 6 months
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | SEL-212A (Low-dose) | SEL-212B (High-dose) | Placebo
Number analyzed (Participants) | 37 | 38 | 37
score on a scale | 7.4 (1.8) | 4.8 (1.7) | 3.0 (1.8)
Statistical Analysis 1: Comparison: SEL-212A (Low-dose) vs Placebo; Test type: Superiority; p = 0.090, Mixed Models Analysis; LS Mean Difference = 4.5, Standard Error of Mean 2.6
Statistical Analysis 2: Comparison: SEL-212B (High-dose) vs Placebo; Test type: Superiority; p = 0.472, Mixed Models Analysis; LS Mean Difference = 1.8, Standard Error of Mean 2.5

5. Secondary Outcome: Proportion of Participants With at Least Partial Response (PR) (as Best Response) in Overall Tophus Response Evaluation in Participants With Tophi at Baseline
Description: Baseline photographs of the hands and feet of each participant were obtained using a standardized method in all participants together with photographs of up to 2 other representative sites of tophaceous disease. The baseline photographs were assessed by three independent reviewers to prospectively identify sites of tophaceous disease present at the start of treatment. Up to 5 tophi in the photographs were chosen by the reviewers for measurement over the course of therapy. The reviewers assessed the photographs for size of each target tophus using image analysis software. At least PR was defined as at least a 50% decrease in the area of at least one tophus, and includes participants with complete response (CR). Data are presented for the proportion of participants with at least PR (as best response).
Time Frame: Baseline up to 6 months
Population: Intent-to-Treat Set, which included all randomized and dosed participants, including participants with missing outcome measure data that were multiple imputed. Participants were analyzed according to randomized treatment. Here, overall number of participants analyzed = participants with tophi at baseline and evaluable data for the outcome measure.
Measure: Number (97.5% Confidence Interval); unit: proportion of participants
Arm/Group | SEL-212A (Low-dose) | SEL-212B (High-dose) | Placebo
Number analyzed (Participants) | 21 | 22 | 21
proportion of participants | 1.00 [NA to NA] — Confidence intervals could not be calculated as the estimated proportion was exactly 1. | 0.67 [0.61 to 0.73] | 0.42 [0.39 to 0.45]
Statistical Analysis 1: Comparison: SEL-212A (Low-dose) vs Placebo; Test type: Superiority; p = 0.0003, Chi-squared; Difference = 0.58, 97.5% CI 2-sided [0.25 to 0.91]
Statistical Analysis 2: Comparison: SEL-212B (High-dose) vs Placebo; Test type: Superiority; p = 0.1895, Chi-squared; Difference = 0.25, 97.5% CI 2-sided [-0.36 to 0.86]

6. Secondary Outcome: Proportion of Participants Who Achieved and Maintained Reduction of sUA < 6 mg/dL for at Least 80% of the Time During Month 6 in the Subset of Participants With Tophi at Baseline
Description: The number of responders in the subgroup of Intent-to-Treat participants with tophi at baseline divided by the number of Intent-to-Treat participants with tophi at baseline.
Time Frame: Baseline up to 6 months
Population: as for outcome 5
Measure: Number (97.5% Confidence Interval); unit: proportion of participants
Arm/Group | SEL-212A (Low-dose) | SEL-212B (High-dose) | Placebo
Number analyzed (Participants) | 21 | 22 | 21
proportion of participants | 0.50 [0.49 to 0.51] | 0.34 [0.33 to 0.36] | 0.07 [0.05 to 0.08]
Statistical Analysis 1: Comparison: SEL-212A (Low-dose) vs Placebo; Test type: Superiority; p = 0.0035, Chi-squared; Difference = 0.43, 97.5% CI 2-sided [0.14 to 0.72]
Statistical Analysis 2: Comparison: SEL-212B (High-dose) vs Placebo; Test type: Superiority; p = 0.0428, Chi-squared; Difference = 0.28, 97.5% CI 2-sided [-0.02 to 0.57]

7. Secondary Outcome: Change From Baseline to Month 6 in Number of Tender Joints
Description: Tender and/or swollen joints were counted. The following joints were assessed: metacarpophalangeal, proximal interphalangeal, and distal interphalangeal joints of the hands; the metatarsophalangeal and interphalangeal joints of the feet; shoulder, elbow, wrist, knee, ankle, tarsus, sternoclavicular, and acromioclavicular joints.
Time Frame: Baseline, Up to 6 months
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: tender joints
Arm/Group | SEL-212A (Low-dose) | SEL-212B (High-dose) | Placebo
Number analyzed (Participants) | 37 | 38 | 37
tender joints | -2.1 (0.3) | -1.4 (0.3) | -1.9 (0.3)
Statistical Analysis 1: Comparison: SEL-212A (Low-dose) vs Placebo; Test type: Superiority; p = 0.517, Mixed Models Analysis; LS Mean Difference = -0.2, 97.5% CI 2-sided [-1.10 to 0.61]
Statistical Analysis 2: Comparison: SEL-212B (High-dose) vs Placebo; Test type: Superiority; p = 0.230, Mixed Models Analysis; LS Mean Difference = 0.4, 97.5% CI 2-sided [-0.39 to 1.28]

8. Secondary Outcome: Change From Baseline to Month 6 in the Total Score of the Health Assessment Questionnaire Disability Index (HAQ-DI)
Description: The HAQ-DI assesses fine movements of the upper extremity, locomotor activities of the lower extremity, and activities that involve both the upper and lower extremities. It includes 20 items in 8 categories: "activity", "arising", "dressing and grooming", "eating", "grip", "hygiene", "reach" and "walking". Scoring within each section was on a 4-point Likert scale from 0 (without any difficulty) to 3 (unable to do), with higher score showing more disability. The average of the 8 category scores was reported as the HAQ-DI total score on a scale of 0 to 3. A decrease in HAQ-DI score from baseline indicated an improvement in the participant's condition.
Time Frame: Baseline, Up to 6 months
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | SEL-212A (Low-dose) | SEL-212B (High-dose) | Placebo
Number analyzed (Participants) | 37 | 38 | 37
score on a scale | -0.2 (0.1) | 0.0 (0.1) | -0.1 (0.1)
Statistical Analysis 1: Comparison: SEL-212A (Low-dose) vs Placebo; Test type: Superiority; p = 0.250, Mixed Models Analysis; LS Mean Difference = -0.1, 97.5% CI 2-sided [-0.35 to 0.12]
Statistical Analysis 2: Comparison: SEL-212B (High-dose) vs Placebo; Test type: Superiority; p = 0.506, Mixed Models Analysis; LS Mean Difference = 0.1, 97.5% CI 2-sided [-0.16 to 0.29]

9. Secondary Outcome: Incidence of Gout Flare During Treatment Periods 1-6 (Months 1-6)
Description: Gout flare was assessed as part of adverse event (AE) collection. Gout flares were assessed during the Treatment Phase using a validated definition of flares in participants with established gout. A gout flare (per Gaffo et al. 2018) was defined as the fulfillment of at least 3 of the following 4 criteria: 1. Participant-defined gout flare, 2. Pain at rest score of >3 on a 0-10-point numerical rating scale, 3. Presence of at least 1 swollen joint, 4. Presence of at least 1 warm joint. Data are presented for the LS mean incidence per month of gout flares during Treatment Periods 1-6 (Months 1-6). A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Months 1-6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: gout flares/month
Arm/Group | SEL-212A (Low-dose) | SEL-212B (High-dose) | Placebo
Number analyzed (Participants) | 37 | 38 | 37
gout flares/month | 0.2 (0.1) | 0.4 (0.1) | 0.3 (0.1)
Statistical Analysis 1: Comparison: SEL-212A (Low-dose) vs Placebo; Test type: Superiority; p = 0.653, ANOVA; LS Mean Difference = -0.1, 97.5% CI 2-sided [-0.55 to 0.37]
Statistical Analysis 2: Comparison: SEL-212B (High-dose) vs Placebo; Test type: Superiority; p = 0.629, ANOVA; LS Mean Difference = 0.1, 97.5% CI 2-sided [-0.36 to 0.56]

10. Secondary Outcome: Incidence of Gout Flare During Treatment Periods 1-3 (Months 1-3)
Description: Gout flare was assessed as part of adverse event (AE) collection. Gout flares were assessed during the Treatment Phase using a validated definition of flares in participants with established gout. A gout flare (per Gaffo et al. 2018) was defined as the fulfillment of at least 3 of the following 4 criteria: 1. Participant-defined gout flare, 2. Pain at rest score of >3 on a 0-10-point numerical rating scale, 3. Presence of at least 1 swollen joint, 4. Presence of at least 1 warm joint. Data are presented for the LS mean incidence per month of gout flares during Treatment Periods 1-3 (Months 1-3). A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Months 1-3
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: gout flares/month
Arm/Group | SEL-212A (Low-dose) | SEL-212B (High-dose) | Placebo
Number analyzed (Participants) | 37 | 38 | 37
gout flares/month | 0.4 (0.1) | 0.4 (0.1) | 0.3 (0.1)
Statistical Analysis 1: Comparison: SEL-212A (Low-dose) vs Placebo; Treatment Periods 1-3 (Months 1-3); Test type: Superiority; p = 0.731, ANOVA; LS Mean Difference = 0.1, 97.5% CI 2-sided [-0.40 to 0.54]
Statistical Analysis 2: Comparison: SEL-212B (High-dose) vs Placebo; Treatment Periods 1-3 (Month 1-3); Test type: Superiority; p = 0.583, ANOVA; LS Mean Difference = 0.1, 97.5% CI 2-sided [-0.35 to 0.58]

ADVERSE EVENTS:
Time Frame: Day 1 up to approximately 12 months
Description: Safety Set, which included all participants who were administered any amount of study drug. Participants were analyzed according to treatment received.
Arm/Group | SEL-212A (Low-dose) | SEL-212B (High-dose) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/37 | 1/38 | 0/37
Serious Adverse Events (participants affected / at risk) | 10/37 | 5/38 | 2/37
Other Adverse Events (participants affected / at risk) | 31/37 | 29/38 | 27/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SEL-212A (Low-dose) (N=37) | SEL-212B (High-dose) (N=38) | Placebo (N=37)
Pneumonia (Infections and infestations) | 1 | 1 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0
Periodontitis (Infections and infestations) | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 2 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SEL-212A (Low-dose) (N=37) | SEL-212B (High-dose) (N=38) | Placebo (N=37)
Gout (Metabolism and nutrition disorders) | 23 | 20 | 23
Hypertriglycerideaemia (Metabolism and nutrition disorders) | 3 | 5 | 1
COVID-19 (Infections and infestations) | 6 | 5 | 2
Cellulitis (Infections and infestations) | 1 | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 1
Folliculitis (Infections and infestations) | 1 | 2 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 2 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 4 | 4 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 2
Hypertension (Vascular disorders) | 4 | 1 | 4
Hypotension (Vascular disorders) | 0 | 2 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 3 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Pyrexia (General disorders) | 0 | 3 | 0
Non-cardiac chest pain (General disorders) | 2 | 0 | 0
Peripheral swelling (General disorders) | 2 | 0 | 0
Gouty tophus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Hepatic steatosis (Hepatobiliary disorders) | 2 | 0 | 0
Blood pressure increased (Investigations) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-12-15): https://cdn.clinicaltrials.gov/large-docs/66/NCT04513366/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/66/NCT04513366/SAP_002.pdf